CLINICAL TRIAL: NCT02972112
Title: Ultrashort Cognitive Behavioral Intervention for Tokophobia- A Prospective Randomized Single Blinded Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: TASMC-16-GA-0155-CTIL
Record Dates: First submitted 2016-10-30; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Specific Phobia
MeSH Terms: conditions — Phobia, Specific | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Study group (Active Comparator): will receive 2 sessions of 90 minutes each of a cognitive behavioral protocol for the treatment of Tokophobia administered by a CBT trained midwife.
  Interventions: Behavioral: CBT
- Control group (Sham Comparator): will receive 2 sessions of a delivery preparation course (practice as usual).
  Interventions: Other: Sham

INTERVENTIONS:
Behavioral: CBT — novel cognitive behavioral protocol for the treatment of tokophobia
  Arms: Study group
Other: Sham — standard birth preparation sessions.
  Arms: Control group

SUMMARY:
Women in their 3rd trimester, represent a unique segment of the tokophobic population. In these cases help is needed within a very short and limited period of time. To date, no specific treatment targets this population in order to ameliorate the anxiety and to provide these women and their newborns with better obstetric and psychiatric outcomes. The present study investigates an accessible individual two session intervention conducted by midwives skilled in CBT (cognitive behavioral therapy) . This intervention is designed to enable stronger emotional regulation and increase of their capacity to accept unexpected changes during labor and feelings of control. The investigators expect this psychological adjustment to lead to a better course of delivery, less interventions including caesarian sections, and subjective birth experience.

ELIGIBILITY:
Inclusion Criteria:

1. Hebrew speaking pregnant women week 32 + 0 to 37 + 0
2. fulfilling the criteria for a specific phobia diagnosed by SCID (Structured Clinical Interview for the Diagnostic) in accordance with DSM-V (Diagnostic and Statistical Manual) and the Fear of Vaginal Delivery Questionnaire (FDQ).

Exclusion criteria:

1. Women who suffer from a psychotic disorder, PTSD or suicidal ideation
2. High risk pregnancies
3. Alcoholism or drug abuse and dependence.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Pregnancy-Related Anxiety Questionnaire | In the end of second session of intervention- up to 4 weeks from screening
  a widely used instrument to assess and identify pregnancy-specific anxiety in women

CONTACTS AND LOCATIONS:
Locations (1):
- The Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] O'Connell MA, Khashan AS, Leahy-Warren P, Stewart F, O'Neill SM. Interventions for fear of childbirth including tocophobia. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013321. doi: 10.1002/14651858.CD013321.pub2. PMID 34231203